CLINICAL TRIAL: NCT01583530
Title: A Randomized, Parallel-Group, Open-Label Study to Evaluate the Absolute Bioavailability, Pharmacokinetics, Tolerability and Safety of a High Concentration Formulation of Belimumab (HGS1006), a Fully Human Monoclonal Anti-BLyS Antibody, Administered Subcutaneously to Healthy Subjects
Brief Title: Study of Belimumab Administered Subcutaneously to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGS1006-C1105
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Belimumab; Injections, Subcutaneous; Drug Administration Routes; Injections; Lupus Erythematosus, Systemic; Lupus; SLE; Systemic Lupus Erythematosus; Antibodies; Autoimmune Disease; Biological Therapy; Immune System Diseases; Pharmacokinetics; Biological Availability
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Immune System Diseases | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Belimumab IV 240 mg (Active Comparator)
  Interventions: Biological: Single Dose Group: Belimumab IV 240 mg
- Belimumab SC 2 x 120 mg (Experimental)
  Interventions: Biological: Single Dose Group: Belimumab SC 2 x 120 mg
- Belimumab SC 1 x 240 mg (Experimental)
  Interventions: Biological: Single Dose Group: Belimumab SC 1 x 240 mg
- Belimumab SC 1 x 200 mg (Experimental)
  Interventions: Biological: Single Dose Group: Belimumab SC 1 x 200 mg
- Belimumab SC 2 x 120 mg weekly (Experimental)
  Interventions: Biological: Multiple Dose Group: Belimumab SC 2 x 120 mg weekly
- Belimumab SC 1 x 200 mg weekly (Experimental)
  Interventions: Biological: Multiple Dose Group: Belimumab SC 1 x 200 mg weekly

INTERVENTIONS:
Biological: Single Dose Group: Belimumab IV 240 mg — Belimumab IV 240 mg administered on Day 0
  Other Names: BENLYSTA™
  Arms: Belimumab IV 240 mg
Biological: Single Dose Group: Belimumab SC 2 x 120 mg — Belimumab SC 120 mg x 2 injections (equal to 240 mg) administered immediately one after the other on Day 0
  Other Names: BENLYSTA™
  Arms: Belimumab SC 2 x 120 mg
Biological: Single Dose Group: Belimumab SC 1 x 240 mg — Belimumab SC 240 mg x 1 injection on Day 0
  Other Names: BENLYSTA™
  Arms: Belimumab SC 1 x 240 mg
Biological: Single Dose Group: Belimumab SC 1 x 200 mg — Belimumab SC 200 mg x 1 injection on Day 0
  Other Names: BENLYSTA™
  Arms: Belimumab SC 1 x 200 mg
Biological: Multiple Dose Group: Belimumab SC 2 x 120 mg weekly — Belimumab 120 mg x 2 injections (equal to 240 mg) administered immediately one after the other on Days 0, 7, 14, and 21
  Other Names: BENLYSTA™
  Arms: Belimumab SC 2 x 120 mg weekly
Biological: Multiple Dose Group: Belimumab SC 1 x 200 mg weekly — Belimumab 200 mg x 1 injection administered on Days 0, 7, 14, and 21
  Other Names: BENLYSTA™
  Arms: Belimumab SC 1 x 200 mg weekly

SUMMARY:
The purpose of this study is to measure the amount of belimumab in the blood when given as an injection under the skin (subcutaneously; SC) and to evaluate the safety and tolerability of multiple injections under the skin in healthy subjects.

DETAILED DESCRIPTION:
This study is designed to evaluate the absolute bioavailability, pharmacokinetics, tolerability, and safety of a single dose (groups 1-4) or multiple doses (groups 5-6) of belimumab administered subcutaneously (SC) to healthy subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy subjects defined as no clinically relevant abnormalities identified by a detailed medical history, full physical exam, 12-lead electrocardiogram (ECG), and clinical laboratory tests.
* Body weight between 45 to 120 kg (99 to 264 lbs).
* Must agree to use effective contraception throughout the study and for 14 weeks after administration of belimumab.
* Have the ability to understand the requirements of the study, provide written informed consent, and comply with the study protocol procedures.

Key Exclusion Criteria:

* Pregnant or nursing.
* Test positive for drugs or alcohol or have had a drug or alcohol dependence within the past year.
* Have used any prescription medicines within the past 30 days or herbal/botanical supplements within the past 7 days or anticipate use during the study. May use prescription contraceptives, hormone replacement therapy, and over-the-counter medicines such as antihistamines or nutritional support such as vitamins, minerals, or amino acids.
* Have received a live vaccine within the past 30 days or anticipate receipt of a live vaccine during the study and within 4 months after last injection of belimumab.
* Have a history of an allergic or anaphylactic reaction to drugs, food, or insect bite or sting requiring medical intervention.
* Have a history of allergic reaction to contrast agents or biological medicines.
* Have participated in a clinical trial and received an experimental medicine within the past 60 days.
* Have received treatment with a B cell targeted therapy at any time.
* Have required management of an infection within the past 14 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - Daytona Beach, Florida
  - Evansville, Indiana
  - Dallas, Texas
  - Madison, Wisconsin

REFERENCES:
- [Derived] Gupta SV, Fanget MC, MacLauchlin C, Clausen VA, Li J, Cloutier D, Shen L, Robbie GJ, Mogalian E. Clinical and Preclinical Single-Dose Pharmacokinetics of VIR-2218, an RNAi Therapeutic Targeting HBV Infection. Drugs R D. 2021 Dec;21(4):455-465. doi: 10.1007/s40268-021-00369-w. Epub 2021 Nov 6. PMID 34741731
- [Derived] Zhou X, Lee TI, Zhu M, Ma P. Prediction of Belimumab Pharmacokinetics in Chinese Pediatric Patients with Systemic Lupus Erythematosus. Drugs R D. 2021 Dec;21(4):407-417. doi: 10.1007/s40268-021-00363-2. Epub 2021 Oct 9. PMID 34628605

RESULTS

PARTICIPANT FLOW:
Groups:
- Belimumab IV 240 mg: Belimumab IV 240 mg administered on Day 0
- Belimumab SC 2 x 120 mg: Belimumab SC 120 mg x 2 injections (equal to 240 mg) administered immediately one after the other on Day 0
- Belimumab SC 1 x 240 mg: Belimumab SC 240 mg x 1 injection on Day 0
- Belimumab SC 1 x 200 mg: Belimumab SC 200 mg x 1 injection on Day 0
- Belimumab SC 2 x 120 mg Weekly: Belimumab 120 mg x 2 injections (equal to 240 mg) administered immediately one after the other on Days 0, 7, 14, and 21
- Belimumab SC 1 x 200 mg Weekly: Belimumab 200 mg x 1 injection administered on Days 0, 7, 14, and 21
Period: Overall Study
Arm/Group | Belimumab IV 240 mg | Belimumab SC 2 x 120 mg | Belimumab SC 1 x 240 mg | Belimumab SC 1 x 200 mg | Belimumab SC 2 x 120 mg Weekly | Belimumab SC 1 x 200 mg Weekly
Started | 19 | 20 | 20 | 19 | 20 | 20
Completed | 19 | 17 | 20 | 18 | 15 | 17
Not Completed | 0 | 3 | 0 | 1 | 5 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Lack of compliance | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belimumab IV 240 mg | Belimumab SC 2 x 120 mg | Belimumab SC 1 x 240 mg | Belimumab SC 1 x 200 mg | Belimumab SC 2 x 120 mg Weekly | Belimumab SC 1 x 200 mg Weekly | Total
Number analyzed (Participants) | 19 | 20 | 20 | 19 | 20 | 20 | 118
Age Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.1) | 33.4 (11.4) | 35.2 (12.1) | 36.1 (9.4) | 33.7 (9.5) | 37.4 (9.7) | 35.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 11 | 8 | 11 | 10 | 65
  Male | 7 | 7 | 9 | 11 | 9 | 10 | 53
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 20 | 19 | 20 | 20 | 118

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Maximum Serum Drug Concentration (Tmax) Following a Single Dose of Belimumab Given as Intravenous Infusion (IV) or Subcutaneous Injection (SC)
Time Frame: Pre-dose, Post-dose on Days 0, 1, 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, and 70
Population: The pharmacokinetic parameter analysis set included all participants who had received at least 1 dose of belimumab and had serum concentration data available through the Day 28 visit. N (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Belimumab IV 240 mg | Belimumab SC 2 x 120 mg | Belimumab SC 1 x 240 mg | Belimumab SC 1 x 200 mg
Number analyzed (Participants) | 19 | 19 | 18 | 18
days | 0.09 [0.05 to 0.30] | 3.9 [0.9 to 9.8] | 4.9 [2.9 to 13.9] | 5.9 [1.9 to 13.9]

2. Secondary Outcome: Time to Reach Maximum Serum Drug Concentration (Tmax) Following Weekly (x 4) SC Injections of Belimumab
Time Frame: Pre-dose, Post-dose on Days 0, 1, 2, 3, 4, 5, 6, 7, 14, 21, 22, 23, 24, 25, 26, 27, 28, 31, 35, 42, 49, 63, 77, 91, and 119
Population: The pharmacokinetic parameter analysis set included all participants who had received 4 weekly doses of belimumab and had serum concentration data available through 7 weeks from first dose. N (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Belimumab SC 2 x 120 mg Weekly | Belimumab SC 1 x 200 mg Weekly
Number analyzed (Participants) | 17 | 19
days | 5.8 (1.5) | 5.5 (1.2)

3. Primary Outcome: Maximum Serum Drug Concentration (Cmax) Following a Single Dose of Belimumab Given as IV or SC
Time Frame: Pre-dose, Post-dose on Days 0, 1, 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, and 70
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Belimumab IV 240 mg | Belimumab SC 2 x 120 mg | Belimumab SC 1 x 240 mg | Belimumab SC 1 x 200 mg
Number analyzed (Participants) | 19 | 19 | 18 | 18
µg/mL | 86.2 (20.0) | 32.7 (29.0) | 31.6 (27.9) | 24.3 (40.3)

4. Primary Outcome: Area Under the Serum Drug Concentration-time Curve From Time 0 to Infinite Time (AUC0-∞) Following a Single Dose of Belimumab Given as IV or SC
Description: AUC (0-∞) = Area under the serum drug concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-last) plus C (last)/λz. C (last) is the last measurable concentration. λz was determined by linear regression (r2 ≥ 0.8) with uniform weighting of all data in the terminal linear portion of the log-transformed drug concentration-time profile.
Time Frame: Pre-dose, Post-dose on Days 0, 1, 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, and 70
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg∙day/mL
Arm/Group | Belimumab IV 240 mg | Belimumab SC 2 x 120 mg | Belimumab SC 1 x 240 mg | Belimumab SC 1 x 200 mg
Number analyzed (Participants) | 19 | 19 | 18 | 18
µg∙day/mL | 1030 (32.1) | 788 (36.1) | 812 (36.2) | 612 (37.9)

5. Primary Outcome: Terminal Elimination Half-life (t1/2,Term) Following a Single Dose of Belimumab Given as IV or SC
Description: Terminal elimination half-life is the time measured for the serum drug concentration of belimumab to decrease by one half.
Time Frame: Pre-dose, Post-dose on Days 0, 1, 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, and 70
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Belimumab IV 240 mg | Belimumab SC 2 x 120 mg | Belimumab SC 1 x 240 mg | Belimumab SC 1 x 200 mg
Number analyzed (Participants) | 19 | 19 | 18 | 18
days | 18.2 (6.3) | 15.9 (5.3) | 18.2 (6.0) | 16.0 (5.1)

6. Primary Outcome: Absolute Bioavailability of a Single Dose of Belimumab Given as IV or SC
Description: Bioavailability (F) is a measurement of the rate and extent to which a drug reaches the systemic circulation. The bioavailability of belimumab administered by IV is compared to the bioavailability of belimumab administered via single-SC injection.
Time Frame: Pre-dose, Post-dose on Days 0, 1, 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, and 70
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: percentage bioavailability
Arm/Group | Belimumab IV 240 mg | Belimumab SC 2 x 120 mg | Belimumab SC 1 x 240 mg | Belimumab SC 1 x 200 mg
Number analyzed (Participants) | 19 | 19 | 18 | 18
percentage bioavailability | NA [NA to NA] — By definition, when a medication is administered IV, its bioavailability is 100%. | 76.1 [64.5 to 89.9] | 81.8 [70.1 to 95.5] | 73.5 [59.7 to 90.5]

7. Secondary Outcome: Maximum Serum Drug Concentration (Cmax) Following Weekly (x 4) SC Injections of Belimumab
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Belimumab SC x 1 200 mg Weekly: Belimumab 200 mg x 1 injection administered on Days 0, 7, 14, and 21
Arm/Group | Belimumab SC 2 x 120 mg Weekly | Belimumab SC x 1 200 mg Weekly
Number analyzed (Participants) | 17 | 19
µg/mL | 21.6 (23.2) | 19.5 (25.1)

8. Secondary Outcome: Area Under the Serum Drug Concentration-time Curve From Time 0 to Infinite Time (AUC0-∞) Following Weekly (x 4) SC Injections of Belimumab
Description: as for outcome 4
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg∙day/mL
Arm/Group | Belimumab SC 2 x 120 mg Weekly | Belimumab SC 1 x 200 mg Weekly
Number analyzed (Participants) | 17 | 19
µg∙day/mL | 763 (29.8) | 661 (31.2)

9. Secondary Outcome: Terminal Elimination Half-life (t1/2,Term) Following Weekly (x 4) SC Injections of Belimumab
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Belimumab SC 2 x 120 mg Weekly | Belimumab SC 1 x 200 mg Weekly
Number analyzed (Participants) | 17 | 19
days | 20.3 (5.2) | 19.8 (4.9)

10. Secondary Outcome: Absolute Bioavailability of Weekly (x 4) SC Injections of Belimumab
Description: Bioavailability (F) is a measurement of the rate and extent to which a drug reaches the systemic circulation. The bioavailability following weekly (x 4) SC injections of belimumab was calculated by comparing the bioavailability of belimumab administered IV to the bioavailability of belimumab administered via 4 weekly SC injections.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (90% Confidence Interval); unit: percentage bioavailability
Arm/Group | Belimumab SC 2 x 120 mg Weekly | Belimumab SC 1 x 200 mg Weekly
Number analyzed (Participants) | 17 | 19
percentage bioavailability | 74.7 [62.6 to 89.1] | 77.9 [67.0 to 90.6]

11. Secondary Outcome: Number of Participants Who Experienced Adverse Events
Description: Includes AEs reported in participants from the first dose of belimumab throughout the study through Day 70/Exit (single dose groups) or Day 119/Exit (multiple dose groups).
Time Frame: Up to Day 119
Population: Analyses were performed on the as-treated population, defined as the set of all participants who received at least 1 partial or full dose of treatment with the assignment to treatment group that was based on the actual treatment administered to the participants.
Measure: Number; unit: participants
Arm/Group | Belimumab IV 240 mg | Belimumab SC 2 x 120 mg | Belimumab SC 1 x 240 mg | Belimumab SC 1 x 200 mg | Belimumab SC 2 x 120 mg Weekly | Belimumab SC 1 x 200 mg Weekly
Number analyzed (Participants) | 19 | 20 | 20 | 19 | 20 | 20
participants
  At least 1 AE | 14 | 11 | 16 | 14 | 18 | 19
  At least 1 serious AE | 0 | 0 | 0 | 0 | 1 | 1
  An AE resulting in death | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to Day 119
Description: Includes AEs reported in participants from the first dose of belimumab throughout the study through Day 70/Exit (single dose groups) or Day 119/Exit (multiple dose groups).
Arm/Group | Belimumab IV 240 mg | Belimumab SC 2 x 120 mg | Belimumab SC 1 x 240 mg | Belimumab SC 1 x 200 mg | Belimumab SC 2 x 120 mg Weekly | Belimumab SC 1 x 200 mg Weekly
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/20 | 0/19 | 1/20 | 1/20
Other Adverse Events (participants affected / at risk) | 14/19 | 11/20 | 16/20 | 14/19 | 17/20 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab IV 240 mg (N=19) | Belimumab SC 2 x 120 mg (N=20) | Belimumab SC 1 x 240 mg (N=20) | Belimumab SC 1 x 200 mg (N=19) | Belimumab SC 2 x 120 mg Weekly (N=20) | Belimumab SC 1 x 200 mg Weekly (N=20)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab IV 240 mg (N=19) | Belimumab SC 2 x 120 mg (N=20) | Belimumab SC 1 x 240 mg (N=20) | Belimumab SC 1 x 200 mg (N=19) | Belimumab SC 2 x 120 mg Weekly (N=20) | Belimumab SC 1 x 200 mg Weekly (N=20)
External ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 3 | 1 | 1 | 3
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 3 | 2
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site oedema (General disorders) | 0 | 0 | 3 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 3 | 9 | 8 | 14 | 14
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site scab (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 3
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster infection neurological (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 2 | 1 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Splinter (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Lymph node palpable (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 3 | 3 | 0 | 5 | 6 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sleep talking (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0
Ovulation pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 4
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multi-center trials, no investigator will be authorized to publish study results from an individual center until the earlier of the multi-center trial results are published or 12 months after the end or termination of the multi-center trial at all sites. All manuscripts and abstracts must be submitted to the sponsor for review at least 30 days prior to submission for publication or for presentation at a scientific meeting. The sponsor may delay publication for up to 3 months.